CLINICAL TRIAL: NCT03278678
Title: Nutritional Screening in Community Living Older Individuals at High Risk of Hospital Admission.
Brief Title: Nutritional Screening in Older Individuals
Status: Completed | Type: Observational
Sponsor: Sanjuan, Silvia Forcano, M.D. (Individual)
Collaborators: Ministerio de Sanidad, Servicios Sociales e Igualdad (Other Government)
Responsible Party: Principal Investigator, Silvia Forcano Sanjuan, Principal Investigator, Sanjuan, Silvia Forcano, M.D.
Other Study IDs: SanjuanS
Record Dates: First submitted 2017-09-06; First posted 2017-09-12 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Malnourished
Keywords: Nutritional screening MNA-SF malnutrition Case Management
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Hospital-based case management programs and home hospitalization services following the risk stratification model of Kaiser Permanente and Kings Fund select an estimated 5% of older individuals living in the community who are at high risk of hospitalization and adverse outcomes. The objective of these services is to avoid deterioration and hospital admissions or visits to the emergency services by regular follow-up, proactive home visits and support of self-care . The prevalence of malnutrition in patients selected using this model of care is unknown.

DETAILED DESCRIPTION:
The aim of this study was to estimate the prevalence of malnutrition, using the MNA, in this high-risk community living population, and to explore risk factors that could identify subgroups of individuals at higher risk.

This study was performed in individuals included in a Case Management (CM) Program lead by the Telemedicine Unit of a tertiary university hospital in Valencia. Patients admitted to the hospital with two or more hospital admissions for medical reasons in the previous year are detected by a computerized system and included in the program, an integrated care intervention developed for patients with complex multimorbidity using patient-centred education activities and integrated care interventions, with the support of a Hospital at Home Unit (HHU). Telephone follow-ups by case manager nurses are focused on identifying problems and detecting disease exacerbations. The main aim of this program is to avoid hospital admissions and reduce the number of visits to emergency services

ELIGIBILITY:
Inclusion Criteria:

* Patients included at Case Management Program for complex chronic condition
* Must be able to answer questions on the telephone

Exclusion Criteria:

* Subjects with no telephone,
* Subjects unable to determine their usual weight
* End-of-life clinical situation

Ages: 65 Years to 105 Years | Sex: All
Age Groups: Older Adult
Study Population: The final sample size was of 791 subjects.
  The baseline characteristics were:
  Mean age (years): 79.9 +/- 10.86 Female : 397 (50.2%) Mean Body Mass Index : 27.6 +/- 5.75
Sampling Method: Probability Sample
Enrollment: 791 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
prevalence of malnutrition | 2 months
  prevalence of malnutrition by using MNA-SF

SECONDARY OUTCOMES:
sexBMI | 2 months
  male or female, average age, BMI
age | 2 months
  average age in years
BMI | 2 months
  body mass index in Kg / m^2

OTHER OUTCOMES:
Risk factors of malnutrition | 2 months
  feeding route, use of dental prosthesis, dysphagia, consistency of foods, specific diets, oral nutritional supplements, patient group, polypharmacy, history of falls, dementia, presence of musculoskeletal, cerebrovascular, gastrointestinal or oncological disease, multimorbidity